CLINICAL TRIAL: NCT02846727
Title: Using Fluorescence Angiography to Detect Occult Shock
Status: Withdrawn | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1509016441
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Hypoperfusion
Keywords: Hypoperfusion; Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis Group: This group will consist of surgical intensive care patients with diagnosis of sepsis, severe sepsis, or septic shock.
  Interventions: Device: skin perfusion image
- Control Group: This group will consist of patients that serve as controls who do not have diagnosis of sepsis, severe sepsis, or septic shock.
  Interventions: Device: skin perfusion image

INTERVENTIONS:
Device: skin perfusion image — Upon enrollment following written, informed consent, the patient will receive an injection of 7.5 mg of Indocyanine Green (ICG) intravenously (Dilute 25 mg of Indocyanine Green (ICG) with 10 cc of solvent to achieve a 2.5 mg/cc concentration.) Following injection, Novadaq's LUNA™ fluorescence angiography system will be utilized to map a standard skin perfusion image (SPI) over the upper extremities and anterior chest wall.

SUMMARY:
The purpose of this study is to determine if fluorescence angiography can detect occult shock (hypoperfusion).

DETAILED DESCRIPTION:
Hypoperfusion may be multifactorial, due to hemorrhage, shock or other disease processes resulting in either capillary leak into the interstitium or profound vasodilatation. Currently, diagnosis of hypoperfusion depends on indirect markers of perfusion such as lactate, blood pressure, creatinine, urine output, and mental status. These are all late signs of hypoperfusion as they are precursors to impending system failure. In this study, the focus will be on one of the most common causes of hypoperfusion in the surgical population; sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis arm inclusion criteria:
* Diagnosis of severe sepsis and septic shock.
* Sepsis is defined as at least two of the following signs and symptoms (SIRS) that are both present and new to the patient and suspicion of new infection:

  * Hyperthermia >38.3°C or Hypothermia <36°C
  * Tachycardia >90 bpm
  * Tachypnea >20 bpm
  * Leukocytosis (>12,000 μL-1) or Leukopenia (<4,000 μL-1) or >10% bands.
  * Hyperglycemia (>120 mg/dl) in the absence of diabetes.
  * Severe sepsis includes SIRS and at least one of the following signs of hypoperfusion or organ dysfunction that is new and not explained by other known etiology of organ dysfunction:
  * Hypotension (<90/60 or MAP <65)
  * Lactate >2
  * Areas of mottled skin or capillary refill >3 seconds
  * Creatinine >2.0 mg/dl
  * Disseminated intravascular coagulation (DIC), Platelet count <100,000
  * Acute renal failure or urine output <0.5 ml/kg/hr for at least 2 hours
* Hepatic dysfunction as evidenced by:

  * Bilirubin >2 or INR >1.5
  * Cardiac dysfunction
  * Acute lung injury or ARDS
* Control arm inclusion criteria:

  * Do not have diagnosis of sepsis, severe sepsis, or septic shock
  * Are not on vasopressors
  * Are normo-thermic

Exclusion Criteria:

* Sepsis arm exclusion criteria:

  * Pregnant
  * Iodide allergy
  * Burns
* Control arm exclusion criteria:

  * Pregnant
  * Iodide allergy
  * Burns
  * Individuals for whom a surrogate decision maker is not available, or is not able to consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients who are 1) primarily assigned to the Division of General Surgery, Trauma, and Surgical Critical Care and 2) admitted to the surgical intensive care units will be screened for eligibility based on enrollment criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Skin Perfusion Value | Up to 6 hours
  We aim to obtain a SPI within 6 hours of enrollment. Skin perfusion images produced by LUNA have computerized, graded quantification of fluorescein intensity (values 0-256). The mean score will be used to compare Sepsis and Control arms.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Pei, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided